CLINICAL TRIAL: NCT07172399
Title: Prevalence and Factors Associated With Pre-hypertension Among Children and Adolescent With Type 1 Diabetes Mellitus
Brief Title: Factors Associated With Pre-hypertension Among Children With Type 1 Diabetes Mellitus
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Ibrahim, aya ibrahim, Sohag University
Other Study IDs: Soh-Med--25-7-6MS
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: blood sampling — blood samples will be taken to discover if there is hyperlipedemia,hyperthrodism or acute kidney injury
Other: • BP will be measured using a calibrated, automated oscillometric device suitable for pediatric use. — All the study participants will be examined for assessment of the height and weight using calibrated equipment, Body Mass Index ,blood pressure will be measured.

SUMMARY:
blood pressure of diabetic patients will be measured

DETAILED DESCRIPTION:
All the study participants will be examined for assessment of the height and weight using calibrated equipment, Body Mass Index (BMI) calculated and plotted against percentiles,Blood Pressure (BP) Measurement:

* BP will be measured using a calibrated, automated oscillometric device suitable for pediatric use.
* Appropriate cuff size will be used based on mid-arm circumference.
* Blood pressure will be measured in the non-dominant arm.
* BP will be measured three times on at least two different occasions, after 5 minutes of rest, in a seated position.
* The average of the readings will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 6 - 18 years, diagnosed with T1DM for at least 1 year and attending the Pediatric diabetes clinic at Sohag University Hospital will be included as cases.

Exclusion Criteria:

Children and adolescents with T1DM associated with autoimmune hypothyroidism or celiac disease and those who had received any form of corticosteroids therapy for any reason in the last 6 months will be excluded.

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: cildren from 6 to 18 year old
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-26 (Actual); Primary Completion 2026-07-25 (Estimated); Study Completion 2026-08-05 (Estimated)

PRIMARY OUTCOMES:
blood pressure | one year
  * BP will be measured using a calibrated, automated oscillometric device suitable for pediatric use.
  * Appropriate cuff size will be used based on mid-arm circumference.
  * Blood pressure will be measured in the non-dominant arm.
  * BP will be measured three times on at least two different occasions, after 5 minutes of rest, in a seated position.
  * The average of the readings will be recorded
  * BP will be measured using a calibrated, automated oscillometric device suitable for pediatric use.
  * Appropriate cuff size will be used based on mid-arm circumference.
  * Blood pressure will be measured in the non-dominant arm.
  * BP will be measured three times on at least two different occasions, after 5 minutes of rest, in a seated position.
  * The average of the readings will be recorded
  * BP will be measured using a calibrated, automated oscillometric device suitable for pediatric

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided